CLINICAL TRIAL: NCT04973657
Title: Phase 1b, Multi-center, Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Safety, Tolerability, PD and PK of VK0214, in Subjects With the Adrenomyeloneuropathy Form (AMN) of X-linked Adrenoleukodystrophy (X-ALD)
Brief Title: A Study to Assess the Pharmacodynamics of VK0214 in Male Subjects With AMN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viking Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: VK0214-102
Record Dates: First submitted 2021-06-28; First posted 2021-07-22 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Adrenomyeloneuropathy Form (AMN) of X-linked Adrenoleukodystrophy (X-ALD)
Keywords: AMN, XALD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VK0214 Active 20mg (Experimental): 20mg QD
  Interventions: Drug: VK0214
- VK0214 Active 40mg (Experimental): 40mg QD
  Interventions: Drug: VK0214
- Placebo (Placebo Comparator): Placebo QD
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VK0214 — API in capsule
  Arms: VK0214 Active 20mg; VK0214 Active 40mg
Other: Placebo — API in capsule
  Arms: Placebo

SUMMARY:
Subjects will be administered multiple doses of VK0214 in a cohort dose escalation process. A total of up to 36 subjects will be enrolled in the study, into one of three dose cohorts. For each cohort, up to 12 subjects will be randomized to receive VK0214 or placebo in a 3:1 ratio so that there will be a total of up to 9 subjects for each of the active doses and up to 3 subjects dosed with placebo in each cohort.

DETAILED DESCRIPTION:
The first part of VK0214-102 will include the first 2 dose cohorts and placebo, which will be dosed in parallel (up to N=24). The first 2 doses used in these cohorts will be 20 mg QD and 40 mg QD for 28 days. A Dose Level Review Team (DLRT) meeting will be held at the end of the first 2 parallel doses.

The DLRT will review safety, tolerability, and preliminary efficacy data from cohort 1 and 2. If the data analyzed show that the first 2 doses are safe and well tolerated the DLRT may make a recommendation for proceeding to commence dosing in the third dose cohort.

Based upon outcomes in Cohorts 1 and 2, the sponsor may decide to include a third dose cohort. Before screening may be initiated in Cohort 3, data to support dosing in this cohort will be submitted to the FDA, together with the amended protocol and the dosing recommendation of the DLRT.

ELIGIBILITY:
Inclusion Criteria:

* Provide a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study and is willing and able to participate.
* Have diagnosis of X-linked adrenoleukodystrophy (X-ALD) by genetic testing and elevated VLCFAs.
* Present clinical features of AMN, or adrenal insufficiency.
* Subjects must be 18 years of age and older.

Exclusion Criteria:

* Have the cerebral form of X-ALD, based on medical records, or based on MRI performed within the last 12 months or MRI at screening
* Have been treated with any drug targeting TRβ or with any drug being tested as therapy for X-ALD AMN form within the past 30 days before screening
* History or presence of clinically significant acute or unstable hepatic, renal, gastrointestinal, pulmonary, immunological, endocrine, diabetes, hematological or oncological that in the opinion of the investigator would pose a significant risk for the subject
* Subject has untreated primary adrenal insufficiency based on morning plasma cortisol and ACTH at screening
* Lorenzo's Oil. Currently taking Lorenzo's Oil or erucic acid containing product, or other lipid lowering agent known to effect VLCFA levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and treatment-emergent serious AEs (TESAEs) | 28 days
  Evaluate the safety and tolerability of multiple oral doses of VK0214 in subjects with AMN

SECONDARY OUTCOMES:
Evaluate the Pharmacokinetics of VK0214 | 28 days
  Pharmacokinetic profile of VK0214 by measuring Peak Plasma Concentration (Cmax)

OTHER OUTCOMES:
Evaluate plasma VLCFAs changes | 28 days
  Evaluate the efficacy of VK0214 on lowering plasma levels of VLCFAs in subjects with AMN

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Viking Clinical Site 203, Palo Alto, California
  - Viking Clinical Site 207, Gainesville, Florida
  - Viking Clinical Site 201, Baltimore, Maryland
  - Viking Clinical Site 205, Seattle, Washington
- France (2):
  - Viking Clinical Site 214, Bordeaux
  - Viking Clinical Site 215, Montpellier
- Viking Clinical Site 209, Leipzig, Germany
- Viking Clinical Site 210, Milan, Italy
- Viking Clinical Site 212, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No